CLINICAL TRIAL: NCT02297971
Title: Assessment of Coagulation and Thrombocyte Function After Termination of Ticagrelor in Patients Who Have Previously Undergone PCI Procedures and Insertion of Coronary Stents
Brief Title: Assessment of Coagulation and Thrombocyte Function After Termination of Ticagrelor
Acronym: BRILIQUE
Status: Completed | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Other Study IDs: 2013/001
Record Dates: First submitted 2014-11-18; First posted 2014-11-21 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: PCI; Coronary Stents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for analysis of complement, coagulation factors and other biochemical markers
Oversight: Data Monitoring Committee: Yes

SUMMARY:
When ticagrelor should be discontinued prior to elective surgery is unclear. The risks of bleeding when it is continued peri-operatively have to be weighed against the risk of coronary artery thrombosis when stopped. This study aims to assess coagulation and thrombocyte function every other day in patients who are taking ticagrelor after coronary artery stents and discontinue therapy at the end of one year.

DETAILED DESCRIPTION:
Patients who have an acute coronary syndrome are today often treated by percutaneous coronary intervention (PCI) and insertion of one or several coronary stents. Subsequently, these patients are treated with oral anti-platelet (OAP) drugs, usually a combination of acetyl salicylic acid (aspirin) and clopidogrel/ticagrelor. Although aspirin is continued for a life-long period, clopidogrel/ticagrelor are used for a variable period of time, often from 3 months - 1 year after PCI, depending on the type of stent. Interventional elective non-cardiac surgery during the time of clopidogrel/ticagrelor therapy is not recommended except for life-threatening (acute surgery) or life-prolonging (cancer surgery) procedures. Specifically for life-prolonging procedures, surgery can be planned, and therefore the question often arises as to when OAPs should be terminated prior to planned surgery. This decision rests on balancing the risks of bleeding (when continued) or coronary stent thrombosis (when stopped). Certainly, because of the small risk of severe bleeding when using aspirin, this drug should be continued throughout the perioperative period in patients with coronary stents. However, continuing clopidogrel/ticagrelor is more controversial since severe perioperative bleeding is difficult to reverse in these patients. Therefore, surgeons would normally discontinue clopidogrel/ticagrelor prior to surgery, specifically when the potential for bleeding is high, and the consequences major. The exact duration for which these drugs should be discontinued remains unclear and, depending on the drug used, a period of 3 - 5 days is generally recommended, based on the pharmacokinetics and dynamics of clopidogrel/ticagrelor in otherwise healthy patients.

This study was done to better understand coagulation and thrombocyte function immediately before discontinuation of ticagrelor and at regular intervals after termination, in patients who have previously undergone PCI, have coronary stents, are taking ticagrelor but discontinue it after one-year of therapy in accordance with hospital routines. No surgical intervention was planned in these patients after termination of ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are on the Cardiology Clinic's database at the University Hospital, Örebro and shall terminate ticagrelor after one year following PCI and stent placement would be identified and offered to take part in this study.

Exclusion Criteria:

- Non-responders (not partial responders) to ticagrelor would be excluded from the study. Additionally, patients who are either taking NSAID's regularly or during the last 2 weeks prior to study start would also be excluded as those who have language or cognitive limitations.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have previously had a coronary artery syndrome treated by PCI and stent placement and who are taking the oral anti platelet drugs aspirin and ticagrelor would be included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Platelet aggregometry | 0 - 10 days
  Platelet aggregometry using Multiplate assay would be done prior to termination of ticagrelor treatment and thereafter every other day of 10 days.

SECONDARY OUTCOMES:
Thromboelstography | 0-10 days
  Thromboelastography would be performed prior to termination of ticagrelor treatment and thereafter every other day of 10 days.
Coagulation function tests | 0-10 days
  Coagulation function would be performed on alternate days starting before termination of ticagrelor.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gupta, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- University Hospital, Örebro, Sweden